CLINICAL TRIAL: NCT03279614
Title: Phase II Study of SOX as the Seconde Line Chemotherapy in Advanced or Metastatic Neuroendocrine Carcinoma
Brief Title: Study to Evaluate the Efficiency of SOX as Seconde-line Chemotherapy in Neuroendocrine Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, MD, Professor, Chief of Department of GI Oncology, Peking University Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOX-2
Record Dates: First submitted 2017-09-10; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Neuroendocrine Carcinoma
Keywords: ORR; OS; PFS; safety
MeSH Terms: conditions — Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOX (Experimental): OXA：130mg/m2 ，iv drip for 180min d1, S-1 40-60mg p.o. bid d1-14, q3W
  Interventions: Drug: SOX

INTERVENTIONS:
Drug: SOX — OXA：130mg/m2 ，iv drip for 180min d1, S-1 40-60mg p.o. bid d1-14, q3W

SUMMARY:
Currently, there is no standard second line treatment for patients with neuroendocrine carcinoma. SOX regimen has shown promising in previous study. The study was designed to confirm thet SOX regimen can be used as a second-line regimen for patients with advanced or metastatic neuroendocrine carcinoma who have progressed after first-line chemotherapy with platinum based regimen.

ELIGIBILITY:
Inclusion Criteria:

1. sign written informed consent form
2. age ≥ 18 years
3. pathologically confirmed poorly-differentiated neuroendocrine carcinoma, G3(Ki67>20%);
4. No prior antitumor treatment with OXA, progress after first line chemotherapy with platinum-based regimen. For recurrent patients after radical surgery, platinum-based adjuvant chemotherapy should beyond 6 months prior to randomization;
5. At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions);
6. Screening laboratory values must meet the following criteria (within past 7 days): hemoglobin ≥ 9.0 g/dL; neutrophils ≥ 1500 cells/ μL; platelets ≥ 100 x 10^3/ μL; total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1╳ULN;
7. KPS ≥ 70;
8. Predicted survival >=3 months;
9. Negative serum or urine pregnant test within 7 days prior to randomization for child-bearing age women;
10. Sexually active males or females willing to practice contraception during the study until 30 days after end of study.

Exclusion Criteria:

1. Hypersensitivity to OXA,5-HT3 receptor antagonists;
2. Prior antitumor therapy (including corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
3. Received surgery within past 4 weeks, or have not recovered from surgery;
4. Severe diarrhea;
5. Concurrent severe infection；
6. Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including severe liver disease (active hepatitis, cirrhosis), uncontrolled diabetes or hypertension, or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm);
7. Prior long term steroid therapy (excluding short term steroid treatment which is completed prior to > 2 weeks of study enrollment)；
8. Meningeal carcinomatosis;
9. Patients with central nervous system(CNS) disorder or peripheral nervous system disorder or psychiatric disease；
10. Known history of uncontrolled or symptomatic angina, uncontrolled arrhythmias and hypertension, or congestive heart failure, or cardiac infarction within 6 months prior to study enrollment, or cardiac insufficiency；
11. Pregnant or nursing, or sexually active males or females refuse to practice contraception during the study until 30 days after end of study;
12. History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, are eligible；
13. Person with no capacity (legally) or inappropriate to continue study treatment for ethics/medical reasons；
14. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  CT/MRI will be performed every 2 cycles of treatment for efficacy evaluation by RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival | baseline, every 8 weeks up to 1 year after last patient first treatment
  Progression-free survival is defined as the time from the date of first dose to the date of the first documented radiological progression or death due to any cause
Overall survival | baseline, every 8 weeks up to 1 year after last patient first treatment
  Overall survival is defined as the time from date of start of treatment to date of death due to any cause
Incidence of Treatment-related Adverse Events （Safety and Tolerability） | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No